CLINICAL TRIAL: NCT02570191
Title: An Open-label, Multicenter, National, Not-randomized Study to Evaluate Efficacy and Safety of Peginterferon Alfa-2a (40 KD) (PEGASYS) in Patients With HBeAg-negative Chronic Hepatitis B
Brief Title: A Study of PEGASYS (Peginterferon Alfa-2a [40KD]) in Patients With Hepatitis B e Antigen (HBeAg)-Negative Chronic Hepatitis B Virus (HBV)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML18092
Record Dates: First submitted 2015-10-05; First posted 2015-10-07 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a

ARMS (1):
- Peginterferon alfa-2a (Experimental): Participants received 180 micrograms (uG) of Pegasys (0.5 milliliter [mL] solution) once a week subcutaneously for 48 weeks.
  Interventions: Drug: Peginterferon alfa-2a

INTERVENTIONS:
Drug: Peginterferon alfa-2a — 180 uG in 0.5 mL solution administered once weekly for 48 weeks
  Other Names: Pegasys

SUMMARY:
This study will evaluate the efficacy, safety, and tolerability of PEGASYS in participants with HBeAg-negative chronic HBV. The anticipated time on study treatment is 48 weeks, and the target sample size is 60 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants 18-70 years of age
* Positive test result for HBsAg for >6 months
* Naive to treatment for HBV
* On liver biopsy, liver disease consistent with chronic HBV, with or without compensated cirrhosis

Exclusion Criteria:

* Co-infection with hepatitis A, C or D, or with Human Immunodeficiency Virus (HIV)
* Decompensated liver disease
* Hepatocellular cancer
* Systemic anti-viral, anti-neoplastic, or immunomodulatory therapy less than or equal to 6 months before study drug
* Medical condition associated with chronic liver disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2004-11; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Efficacy: Hepatitis B Virus - Deoxy ribonucleic acid (HBV-DNA) less than (<)20,000 Copies per milliliter (copies/mL) At End of Follow-Up | 72 Weeks
Alanine Transaminase (ALT) Normalization at the End of Follow-Up | 72 Weeks

SECONDARY OUTCOMES:
Efficacy: Loss of Hepatitis B Virus Antigen ( HBsAg) and Seroconversion at End of Follow-Up | 72 Weeks
Hepatitis B Virus (HBV) DNA Below the Limit of Quantification At the End of Follow-Up | 72 Weeks
HBV DNA Suppression <20000 Copies/mL at the End of Treatment | 48 Weeks
Alanine Transaminase (ALT) Normalization at the End of Treatment | 48 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (4):
- Bulgaria (4):
  - Pleven
  - Plovdiv
  - Sofia
  - Stara Zagora